CLINICAL TRIAL: NCT03311321
Title: Vitamin K to Slow Progression of Cardiovascular Disease Risk in Hemodialysis Patients (Vita-K 'n' CKD Study)
Brief Title: Vitamin K to Slow Progression of Cardiovascular Disease Risk in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Norman Pollock, Associate Professor, Department of Medicine, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 683534
Record Dates: First submitted 2017-10-09; First posted 2017-10-17 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Cardiovascular Diseases; Chronic Kidney Disease Stage 3; Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 5; Vitamin K Deficiency; Hemodialysis
Keywords: Arterial Stiffness; Endothelial Function; Vitamin K
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic; Vitamin K Deficiency | interventions — Vitamin K 2; menaquinone 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-Control (Placebo Comparator): The placebo-control group will take four placebo softgel capsules (similar in taste and appearance to the vitamin K2 supplements) every day for 8 weeks.
  Interventions: Dietary Supplement: Placebo-Control
- Vitamin K2 (360-mcg/d) (Experimental): The experimental group will take four 90-mcg of vitamin K2 (menaquinone-7; 360-mcg) softgel capsules every day for 8 weeks.
  Interventions: Dietary Supplement: Vitamin K2 (menaquinone-7; 360-mcg/d)

INTERVENTIONS:
Dietary Supplement: Vitamin K2 (menaquinone-7; 360-mcg/d) — four 90-mcg vitamin K2 (menaquinone-7) softgel capsules per day for 8 weeks
  Arms: Vitamin K2 (360-mcg/d)
Dietary Supplement: Placebo-Control — four placebo softgel capsules per day for 8 weeks containing no vitamin K2 (menaquinone-7)
  Arms: Placebo-Control

SUMMARY:
The life span of adults with end-stage renal disease is reduced, and cardiovascular disease (CVD) accounts for approximately half the deaths among those undergoing hemodialysis (HD). Vascular calcification is a key process in the development of atherosclerotic and arteriosclerotic CVD, and contributes significantly to the greater mortality rates and CVD events in HD patients. Recently, there has been growing interest in the vitamin K-dependent matrix Gla protein (MGP) and its role in inhibiting vascular calcification. Animal studies have revealed that the vitamin K-dependent protein MGP may reduce the progression of vascular calcification, possibly by means of improving vascular function. The relationship between MGP and vitamin K lies in the fact that inactive matrix Gla protein requires vitamin K to carboxylate it for its activation. Currently, data in HD patients are scant and equivocal on the effects of vitamin K supplementation on CVD risk outcomes. Therefore, the purpose of this 8-week randomized, placebo-controlled, double-blind clinical trial is to determine whether daily vitamin K supplementation can favorably alter measurements of endothelial function and arterial stiffness in HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease Stages 3 to 5
* Receiving hemodialysis treatment for at least 3 months
* Subject understands the study protocol and agrees to comply with it
* Informed consent documents signed by subject

Exclusion Criteria:

* Using vitamin supplements containing vitamin K
* History of metabolic gastrointestinal diseases
* Subjects presenting chronic degenerative and/or inflammatory diseases
* Receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters (salicylates, antibiotics)
* Subjects receiving corticosteroid
* Use of anticoagulants
* History of soy allergy
* Have an unstable medical condition, such as having a life expectancy of less than 6 months in the judgment of the investigator
* Known sensitivity, intolerance, or other adverse response to study drugs which would prevent compliance with study medication
* Subjects who have participated in a clinical study more recently than one month before the current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Flow-Mediated Dilation (FMD) | Change from baseline to 8 weeks
  The FMD test is non-invasive assessment of vascular endothelial function.
Pulse Wave Velocity (PWV) | Change from baseline to 8 weeks
  The PWV test is a non-invasive test of arterial stiffness.

SECONDARY OUTCOMES:
Prothrombin Time | Change from baseline to 8 weeks
  The prothrombin time test is a measurement of clotting time.

CONTACTS AND LOCATIONS:
Overall Officials: Norman K Pollock, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
1. Approximate date of when the data will be shared? 2019-06-01
  2. Where will the data be made available? The de-identified data will be made available for research purposes only by contacting the principal investigator.
  3. Please explain any limits to data sharing that might be required. Even though the final research data will be stripped of identifiers prior to release for sharing, the investigators believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, the principal investigator will make the data available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available on June 1, 2019 for approximately 12 months.
Access Criteria: The principal investigator will make the data available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
URL: http://www.augusta.edu/mcg/dphs/gpi/clinicalresearch.php

REFERENCES:
- [Background] Fain ME, Kapuku GK, Paulson WD, Williams CF, Raed A, Dong Y, Knapen MHJ, Vermeer C, Pollock NK. Inactive Matrix Gla Protein, Arterial Stiffness, and Endothelial Function in African American Hemodialysis Patients. Am J Hypertens. 2018 May 7;31(6):735-741. doi: 10.1093/ajh/hpy049. PMID 29635270
- See also: Principal Investigator - Faculty Profile — https://www.augusta.edu/faculty/directory/view.php?id=NPOLLOCK